CLINICAL TRIAL: NCT07355556
Title: Technology Supported Improvement, Management and Prevention of Accidental Falls in Hospitals
Acronym: TechSIMPAFiH
Status: Not yet recruiting | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: University Hospitals, Leicester (Other); Northern Care Alliance NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 25057
Record Dates: First submitted 2025-11-14; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-10

CONDITIONS: Accidental Falls; Fall Prevention
Keywords: ethnographic case study; contextual enquiry; observation of clinical staff; The use of technology to prevent falls; mixed methods research

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- clinical ward team UHL1: A clinical ward team in a NHS acute care Trust
- clinical ward team UHL2: A clinical ward team in a NHS acute care Trust

SUMMARY:
The student will observe fall prevention systems in practice in 2 different hospitals considering how fall prevention technology influences staff behaviour and patients safety in the context of accidental falls in hospital. Accidental falls in hospital are rare but can be life changing for those that suffer them as they are often frail patients who are already vulnerable. Current research shows little improvement with any interventions tested which leaves patient facing clinicians with few resources to assist in the prevention of falls. The investigator believes this is because the measure of accidental falls in hospital is not sensitive enough to calibrate for the different contexts in which patients fall. The student would posit that it is the context that is most influential and addressing the context may lead to improved measures so progress can be made in finding solutions.

DETAILED DESCRIPTION:
The multi-centre study will involve up to 2 wards on each of the 2 Trust sites. The study wards will be randomly selected from a group of wards that have indicated they are happy to be considered as potential research wards. An ethnographic case study with contextual enquiry design will be used to allow a contextual analysis of fall prevention in practice and consider how staff decisions and behaviour contribute to this. Hierarchical task analysis (HTA) will be utilised to inform this and to identify differences between 'work as imagined' compared to 'work as done' . The study will use observations of the staff in clinical practice using their current system of fall prevention measures assisted by their existing technology and will illustrate outcomes with specific and transparent definitions. Calculations of falls occurring measured with local live data will compare with current standard measurements (Falls/1000 occupied bed days) as calculated with central occupancy data. The ward team, patients and relatives attending the wards will have an opportunity to complete a questionnaire about the use of fall prevention technology advertised in the ward environment on fliers and posters as permitted by policy. Recommendations for future technology design, research and use of technology in fall prevention will be provided on conclusion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Any member of the ward team as defined by the ward manager including students. All healthcare professional groups, ancillary and administrative staff who work on the selected study ward and any temporary staff from agency or other wards who consent to participate.

Exclusion Criteria:

* Any staff under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthcare professionals working as a clinical team in practice
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
To discover how work practice and behaviour adheres or varies from policy | 12 months
  Data will be gathered by observing staff in their usual work environment over a 12 month period to determine how fall prevention practice is shaped by technology. Up to 200 staff will be observed by the researcher on various shifts. Hierarchical task analysis will be used to compare how work varies from the policy/protocol and any workarounds that have been developed (Work as done will be compared to work as imagined). Adherence to policy/protocol or variance from policy/protocol will be recorded and collated as a count of deviations.
To collate evidence of the context of falls in a context log to identify potential contributory factors to accidental falls in hospital. | 12 months
  A thematic analysis of accidental fall incident forms will be undertaken comparing contextual details at the time of the accidental fall to identify common themes. Previously uncollated facts such as the exact location of fall (bedside or bathroom), lighting at the time and ability to alter the lighting (automatic switch on /off versus dimmer switch), footwear (own or provided in hospital) and whether walking aids in place or not etc. These will be compared before the implementation of fall prevention alarms versus after implementation to see if the implementation of fall prevention alarms has impacted on falls in any specific contextual category. This will identify if there is a specific context in which fall prevention alarms prevents falls. This will allow more accurate measurement of success of technology as there may be a specific type of fall that can be prevented by the technology.
To discover how accidental falls are being measured and recorded in hospital by observation and comparing live data measurement against standard data measurement. | 12 months
  The current way of calculating falls/1000 bed days is flawed. Occupancy rate and number of admissions are not considered. The outcome will compare standard falls/1000 OBD's versus a contextual measurement that better represents outcomes. Instead of taking average hospital occupancy data the calculation of the number of falls/1000 occupied bed days will be calculated using actual data from ward level occupancy. If the hospital uses an electronically generated occupancy measurement it can give falsely high measurements of falls on a specific ward as it reports empty beds at midnight. These empty beds at midnight are often an electronic delayed transfer rather than actual empty beds. measurement according to stafff reported figures will be compared.

SECONDARY OUTCOMES:
To identify through thematic analysis using Nvivo 15 task critical attributes and user requirements for future fall prevention technology design | 12 months
  The observation of the use of technology in practice will provide themes where practice is impeded or enhanced by the use of technology. This will be identified by the themes identified during observation of staff. These themes will be analysed and recommendations for future fall prevention alarms will be deduced.
Staff interviews | 12 months
  Staff will be questioned during their shift with 'go along questions' (quick questions in between work tasks) to record their rationale for completing fall prevention tasks in the way they have. Answers will be anonymously recorded to provide themes to be analysed using Nvivo 15.

CONTACTS AND LOCATIONS:
Overall Officials: James Reid, Principal Investigator — University Hospitals, Leicester
Locations (1):
- University Hospitals of Leicester, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided